CLINICAL TRIAL: NCT05680376
Title: Relationship Between Habitual Abortion With Thyroid Hormone Values and Anti-TPO (Anti-thyroid Peroxidase Antibody) Positivity
Brief Title: Thyroid Hormone Values and Anti-thyroid Peroxidase Antibody Positivity in Recurrent Pregnancy Loss
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Büşra Özgen Çeviker, Resident at Family Medicine Department, Zonguldak Bulent Ecevit University
Other Study IDs: 2022/17
Record Dates: First submitted 2022-11-30; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Autoimmune Thyroiditis; Recurrent Miscarriage
Keywords: Thyroid Hormones; Anti Thyroid Peroxidase Antibody; Recurrent pregnancy loss
MeSH Terms: conditions — Thyroiditis, Autoimmune; Abortion, Habitual

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recurrent Pregnancy loss: patients with a diagnosis of recurrent miscarriage
- Healthy Controls: healthy women at same age and similar demographics

SUMMARY:
The aim of this study is to compare the thyroid hormone values and anti-thyroid peroxidase (anti-TPO) levels of women with a diagnosis of recurrent pregnancy loss (RPL) and healthy pregnancies. The primary objective is to find out the relationship between recurrent pregnancy loss with thyroid hormone levels and anti-TPO positivity.

ELIGIBILITY:
Inclusion Criteria:

* women with 2 or more pregnancy loses
* for controls women with least one healthy baby

Exclusion Criteria:

* any other metabolic disease
* women with one miscarriage

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The study was carried out with a total of 103 patients by retrospectively examining the patients who applied to the Gynecology and Obstetrics Clinic of Bülent Ecevit University Faculty of Medicine between 2018-2022
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Anti-thyroid Peroxidase Antibodies | 4 years
  presence of Anti-thyroid Peroxidase Antibodies in both groups
Thyroid Hormone Levels | 4 years
  levels of Thyroid stimulant Hormone, Thyroxin and triiodothyronine levels

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bulent Ecevit University Faculty of Medicine, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No